CLINICAL TRIAL: NCT03482466
Title: A Virtual World/Neurofeedback Real Time Functional MRI Approach to PTSD Treatment
Brief Title: Machine Learning Neurofeedback for PTSD
Acronym: NEUROFPTSD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2588-P
Record Dates: First submitted 2018-03-16; First posted 2018-03-29 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-03

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: 12 PTSD patients will be exposed to the real time functional MRI neurofeedback training. The investigators will assess PTSD symptoms both clinically and with a "take home" wearable device that will collect data on physical activity, heart rate, and sleep patterns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PTSD patients (Experimental): 12 PTSD patients will be recruited to undergo neurofeedback training .
  Interventions: Behavioral: Neurofeedback

INTERVENTIONS:
Behavioral: Neurofeedback — Patients will be inside an MRI machine. They will be trained using real time feedback from brain imaging to learn personal strategies to bring their brain to the CALM state.
  Other Names: Real time fMRI virtual reality training

SUMMARY:
A commonly used therapy for post-traumatic stress disorder (PTSD) that often (but not always) gives good results is "exposure therapy": When the patient (for example, Veterans who have attacks of anxiety when a noise startles them) talks about the trauma that precipitated the PTSD, she or he slowly becomes less sensitive to PTSD. This works only on some patients. The investigators propose to expose PTSD patients to a number of "training" sessions in which they will be in a virtual world (similar to a video game) driving a car through a place resembling Iraq. This will happen inside an MRI machine, and the investigators will obtain brain images while the patient is exploring the "virtual Iraq" environment. The investigators will project on the screen a bar that will let the patient know, in real time, which is the state of her or his brain, from CALM to STRESS. The job of the patient will be to try to come up with personal strategies (breathe slowly, think calming thoughts) to try to bring the bar to CALM. The investigators believe that after a number of sessions, the patient will be able to create personalized mental strategies to bring their brain to CALM state, even in real life. This could become a much stronger way of performing "exposure therapy". Finally, the investigators will use a wearable device (similar to a wristwatch) to be able to study physical activity and sleep patters in PTSD patients through the training, in the hope that the investigators may find a way to objectively study when a patient is doing better.

DETAILED DESCRIPTION:
A Virtual World/Neuro-feedback Real-time Functional MRI Approach to PTSD Treatment

Despite availability of treatment, posttraumatic stress disorder (PTSD) remains a major problem in Veterans, with tremendous impact on patients, their families, and the VHA system. A major therapeutic approach used for Veterans with PTSD is exposure therapy, with beneficial effects in many patients. However, improvements on current therapies are needed.

The overarching hypotheses of this proposal are two-fold. First, that brain activity measured with functional MRI (fMRI) can be used to discern the different brain states of a PTSD patient during a threatening experience vs. during a calm moment, and that patients, aided by neuro-feedback derived from real-time fMRI during a virtual reality experience, can learn to reduce their response by willfully modifying their brain state. Secondly, that the continuous measurement of physical activity, heart rate, and sleep patterns using wearable devices can help in the study of PTSD treatment trajectories.

Investigators will combine virtual worlds, machine learning, real-time fMRI, and neuro-feedback to provide a novel PTSD treatment that the investigators hope will be more effective than current alternatives, at least in certain challenging cases. The investigators will construct a computational model specific for patient+stimulus combination. This is critical as PTSD patients are very heterogeneous.

Aim 1. Use of Virtual World/Neurofeedback with Real-Time fMRI as therapy for PTSD Fifteen PTSD patients recruited at MEDVAMC will be exposed to Virtual Iraq, a virtual world platform in which they will be exposed to war-like scenarios, and to calm scenes where no threat will be present. Brain activity will be collected using fMRI and analyzed with machine learning to discern between both extreme brain states (STRESS vs. CALM). These two states will be used during neurofeedback training: In the following weeks, participants will be exposed to 7 fMRI/Virtual World sessions in which they will be instructed to try to move a gauge to the CALM side by using individual mental strategies (active like concentrating on a particular memory, or passive as it has been shown that neurofeedback does not necessarily need willful effort to work). The stressfulness of the Virtual World will be manipulated by the gauge: when the patient is able to move the bar toward CALM (by bringing the brain toward that state) the stressfulness of the Virtual World will decrease.

Hypothesis 1: PTSD symptoms will decrease as training progresses and patients learn mental strategies to "bring the world" to a CALM state.

Aim 2. Study of wearable technology to assess treatment success in PTSD While there are PTSD measuring tools and the investigators will use them before, during, and after training, in general self-reports are not as robust and reliable as one would like. Thus, it would be beneficial to have more physiological measures of treatment progression for PTSD, and for psychiatry in general. The investigators will use a wearable device similar to a wristwatch that the participant will continuously wear throughout the training.

Hypothesis 2: Data from the wearable device will correlate with self reports and with increased ability to willfully bring the Virtual World to the CALM state during training.

The investigators propose that neurofeedback will give PTSD patients the possibility of discovering personal mental strategies to become calmer. However, this learning does not need to be the result of willful effort, as it has been shown that real time fMRI-related learning can occur without conscious effort. In addition, the investigators postulate that wearable devices will capture physiological data linked to the trajectories during PTSD treatment.

The approach may be too expensive to be routinely used (a careful post-study cost-benefit study may prove otherwise, though). However, if this pilot is successful, it may be possible to use this data to develop less expensive hybrid alternatives to add to exposure therapy, such as using fMRI in combination with EEG to discern between brain states (only one MRI visit needed), and then using only EEG during training.

Preliminary Studies The research in this proposal will build upon the investigators' 4-year research project at UT Austin funded by the Army Research Office. That work greatly extended the utility of 3D Virtual Worlds for use as stimuli for fMRI-based research, and laid the groundwork for individualized therapies and training. It will play a central role in providing neuro-feedback by analyzing brain activity of patients in response to virtual worlds designed to elicit PTSD responses, such as those provided by BRAVEMIND.

fMRI data acquisition samples a volume of brain activity every 2-3 seconds for several minutes as needed. Each sample is a 3D array of voxels that measure the aggregate brain activity for a few million neurons. Conventional fMRI data analysis treats the values from each voxel as separate time series, and performs a linear statistical analysis that relates the stimulus to the measured activity. To deal with the increased complexity of using real-time virtual worlds as a stimulus, the investigators instead used machine learning for analysis. Machine learning based methods can extract complex correlations over many voxels rather than a single voxel. The method involves "training" by feeding example input/output pairs into the algorithm. In the investigators' case, the input is an fMRI time sample and the output, reflecting the stimulus, is a category in which the investigators are interested. The investigators refer to each category as a "brain state", which is the brain activation pattern specified by labeling each time slice with a particular stimulus category.

The investigators were able to achieve accurate performance for detecting brain states in two different experiments. Both used virtual worlds suggestive of Iraqi towns and virtual characters of U.S. Army and native hostile combatants. In the first experiment, the investigators used a passive viewing paradigm in which 1-6 combatants were presented at different locations in a virtual town. Performance averaged across subjects was quite good and far above chance in terms of determining how many combatants (1-6) was the participant seeing at each time. The second experiment used a similar but more complex stimulus that included a specific visual task requiring user reaction. Subjects were asked to rapidly respond via a button press to a weapon being pulled out suddenly by a single hostile combatant within a crowd of 20 characters, half of which were friendly forces. Task difficulty was varied randomly over encounters that lasted 30 sec each. The investigators' machine-learning methods could recognize this brain state dimension with 70%-90% accuracy.

Research Design and Methods Aim 1. Use of Virtual World/Neurofeedback with Real-Time fMRI as therapy for PTSD The investigators will combine virtual worlds, real-time fMRI, machine learning, and neuro-feedback, to provide a novel PTSD treatment that the investigators hope will be more effective than current alternatives. The investigators also anticipate that by examining the brain maps like those above the investigators will gain insight into how PTSD manifests in the brains of different subjects. The stereo audio/visual stimulus will be provided by the BRAVEMIND system. Prior to scanning, each subject will participate in a side-lab therapy session attended by a trained therapist. The investigators will adjust stimulus parameters to provide an appropriately therapeutic range of responses between CALM and STRESSED. Various scenes/scenarios will be available. This range of parameter settings will be captured for subsequent scanning sessions. In the scanner, the virtual-reality stimuli will be delivered using an MR-compatible 3D display. Subjects will provide self-report their level of "STRESSED" anxiety using a five-button MR-compatible response device. This response data and the MRI data from the first two sessions will be used by machine-learning algorithms to build classifiers that can discriminate the subject's responses between CALM - STRESSED at every 1.5 sec time sample. In the following 6 sessions, the subject will be presented with similar but not identical stimuli while receiving feedback from the machine learning. This will enable them to gradually learn how to self-modulate their own brain response toward a calmer reaction. Such self-induced changes will be detected by the fMRI system and will be used to modulate the virtual world to directly reduce the degree of perceived threat; thus, providing the real-time neuro-feedback required by extinction therapy (a "thermometer" will be displayed).

Whole-brain FMRI data will be collected using a 3T Siemens Prisma scanner using SMS acceleration to obtain 2-mm voxel size and TR = 1.5 sec (SMS x3, G = 2, TE = 30 ms, FA = 72 ). Scanning sessions will last ~1 hour, and begin with the collection of localizers and a high-resolution anatomy (MP-RAGE), 1-mm cubic voxels, followed by the collection of fMRI data during virtual-reality stimulus presentation. Each fMRI run will last ~6 min, and 6-8 runs will be collected.

Pitfalls and alternative strategies. The investigators have demonstrated the ability to classify an internal brain dimension with 89% accuracy, but it may not be possible to obtain similar accuracy for the "PTSD" dimension. It may be possible to improve results by including the observed pulse and respiration data as input into the machine learning. Moreover, even if the feedback is unsuccessful, the investigators will still gain insights into the physiology of PTSD from the sensitivity maps that are generated by the machine learning.

Aim 2. Study of wearable technology to assess treatment success in PTSD Physical activity, heart rate, and sleep patterns all play important roles in PTSD. Wearable technology has recently evolved such that the investigators can now constantly measure these three parameters in a non-invasive manner throughout the course of a study. The investigators propose to study self-reported symptoms in conjunction with physical activity, sleep patterns, and heart rate date over 9 weeks. The investigators will use linear regression to study whether CAPS5, PCL, and diary symptoms correlate with activity, sleep, and heart rate patterns during treatment. The investigators hypothesize that in patients in which the treatment is most successful, a) Average HR will decrease more, b) Bouts of high HR during day and night will be less common, c) Average physical activity will increase, d) Physical activity will regularize to more activity during the day and less activity during the night, e) Average time asleep will increase, and f) Sleep patterns will regularize with less awake epochs during the night.

Pitfalls and alternative strategies. It is possible that the data from wearable devices will not correlate with symptom improvement. A likely explanation would be that the error rate of current devices does not allow for correlations to be significant. If that is the case, this approach should be tested again in the future. Another less likely explanation would be that physical activity, heart rate, and sleep quality are not as strongly correlated with PTSD symptoms as the available data suggests. Since this is a small pilot study, data suggesting a trend would point into possible directions to study in the future.

General conclusion The main idea of the study is that the VR will change to a less stressful environment as the brain approaches the state previously defined as CALM. The investigators postulate that over time, patients will learn to consciously bring their brain to CALM state, which will provide them with individualized mental strategies to calm down when a trauma/stress trigger is present.

ELIGIBILITY:
Inclusion Criteria:

* Meet CAPS5 PTSD criteria
* OEF/OIF/OND & PGW Veterans
* Seeking treatment for PTSD

Exclusion Criteria:

* DSM-5 criteria for drug or alcohol abuse or dependence in past 30 days
* History of moderate to severe traumatic brain injury
* Presence of contraindications to MRI
* Current neurological or general medical conditions known to impact cognitive and/or emotional functioning (epilepsy, Parkinson's, etc.)
* Acute psychological instability, schizophrenia, etc.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramiro Salas, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled during 2018, 2019 and 2020. Study enrollment was stopped in March 2020 due to COVID-19 social distancing protocols.
Groups:
- PTSD Patients: Neurofeedback: Patients will be inside an MRI machine. They were trained using real time feedback from brain imaging to learn personal strategies to bring their brain to the CALM state.
Period: Overall Study
Arm/Group | PTSD Patients
Started | 14
Completed (2 of the 14 study participants did not complete the study protocol. These 2 study participants were removed from the study for inappropriate/ uncooperative behavior.) | 12
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: While 14 participants were recruited overall, 2 of the 14 study participants did not complete the study protocol. These 2 study participants were removed from the study for inappropriate/ uncooperative behavior. Thus, 12 study participants are used for the purpose of analysis.
Groups:
- PTSD Patients: Following assessment for eligibility and safety, study participants view an audiovisual stimulus called Bravemind, a virtual-world environment for military members simulating Iraq and Afghanistan. The interaction involves passive view of a virtual town with an appearance similar to those found in Iraq and Afghanistan. Events occur in the stimulus designed to evoke stress, such as smoke, explosions, and/or the appearance of enemy combatants. While viewing this environment, study participants are undergoing an fMRI scan and rating their level of stress on a 1-8 scale. There is no control group for this study.
Arm/Group | PTSD Patients
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.00 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Clinician Administered PTSD Scale for DSM-5 [Mean (Standard Deviation); unit: units on a scale] — The Clinician-Administered PTSD scale for DSM-5 (CAPS-5) produces reliable and valid scores with standard administration. The CAPS-5 should be administered by qualified interviewers with formal training in structured clinical interviewing and differential diagnosis, a thorough understanding of the conceptual basis of PTSD, and detailed knowledge of the features and conventions of the CAPS-5 itself. The CAPS-5 severity ratings are based on symptom frequency/ amount and symptom intensity. Scores range from 0 - 80, with higher scores indicating increased PTSD symptom severity.
  units on a scale | 37.08 (9.19)

OUTCOME MEASURES:

1. Primary Outcome: CAPS-5 PTSD Criteria
Description: Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a 30-item structured interview that can be used to determine: current (past month) diagnosis of PTSD, lifetime diagnosis of PTSD, PTSD symptoms over the past week. Scores range from 0 - 80, with higher scores indicating increased PTSD symptom severity. The full interview takes 45-60 minutes to administer.
  In addition to PTSD symptoms, questions target symptom onset and duration, subjective distress, impact of symptoms on social and occupational functioning, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization). The CAPS-5 produces reliable and valid scores with standard administration. It should be administered by qualified interviewers with formal training in structured clinical interviewing and differential diagnosis, a thorough understanding of the conceptual basis of PTSD, and detailed knowledge of the measure's features and conventions.
Time Frame: 6 weeks
Population: Data cannot be reported : Due to social distancing procedures implemented during the COVID-19 pandemic, only baseline data was collected for study participants. Thus, study participants were not assessed again at 6 weeks as originally planned.
Arm/Group | PTSD Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Wearable Device Data: Heart Rate
Description: The investigators will collect heart rate data from wearable devices. It will be used to study any possible correlations between wearable device results and changes in CAPS5 during the training, regardless of whether the changes in CAPS5 are due to the training or not. Heart rate will be measured over time in beats per minute.
Time Frame: Change from baseline at 6 weeks
Population: Outcomes could not be measured because the protocol was not completed due to unexpected complications including COVID-19. The investigators were unable to obtain the necessary measures. The investigators did not collect any heart rate data.
Arm/Group | PTSD Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Wearable Device Data: Sleep Patterns
Description: The investigators will collect sleep pattern data from wearable devices. It will be used to study any possible correlations between wearable device results and changes in CAPS5 during the training, regardless of whether the changes in CAPS5 are due to the training or not. Sleep patterns will be measured over time in number of wake events per night.
Time Frame: Change from baseline at 6 weeks
Population: This outcome could not be measured because the protocol was not completed due to unexpected complications including COVID-19. The investigators did not collect any sleep data.
Arm/Group | PTSD Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Wearable Device Data: Total Sleep
Description: The investigators will collect total sleep data from wearable devices. It will be used to study any possible correlations between wearable device results and changes in CAPS5 during the training, regardless of whether the changes in CAPS5 are due to the training or not. Total sleep will be measured over time in minutes of sleep per day.
Time Frame: Change from baseline at 6 weeks
Population: as for outcome 3
Arm/Group | PTSD Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- PTSD Neurofeedback: Following assessment for eligibility and safety, study participants view an audiovisual stimulus called Bravemind, a virtual-world environment for military members simulating Iraq and Afghanistan. The interaction involves passive view of a virtual town with an appearance similar to those found in Iraq and Afghanistan. Events occur in the stimulus designed to evoke stress, such as smoke, explosions, and/or the appearance of enemy combatants. While viewing this environment, study participants are undergoing an fMRI scan and rating their level of stress on a 1-8 scale. There is no control group for this study.
Arm/Group | PTSD Neurofeedback
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Due to unforeseen circumstances including COVID-19, we were unable to complete the whole project.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03482466/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03482466/ICF_001.pdf